CLINICAL TRIAL: NCT03854838
Title: A Single Center 、Single Arm Phase I/II Clinical Trial of Intensity-modulated Radiotherapy Combined With Toripalimab in the Treating of Unresectable Locally Recurrent Nasopharyngeal Carcinoma.
Brief Title: IMRT Combined With Toripalimab in Unresectable Locally Recurrent Nasopharyngeal Carcinoma.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Ming-Yuan Chen, principal investigator, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-FXY-020
Record Dates: First submitted 2019-02-24; First posted 2019-02-26 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Nasopharyngeal Carcinoma; Nasopharyngeal Neoplasms; Nasopharyngeal Diseases; Head and Neck Neoplasm
Keywords: toripalimab; IMRT; Intensity-Modulated Radiation Therapy; PD-1
MeSH Terms: conditions — Nasopharyngeal Carcinoma; Nasopharyngeal Neoplasms; Nasopharyngeal Diseases; Head and Neck Neoplasms | interventions — Re-Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Toripalimab +Radiotherapy (Experimental): Radiotherapy, intensity-modulated radiation therapy (IMRT), 60 Gy 2.2Gy per fraction ,5 fractions per week, for 6 weeks. Radiation begun the day after the first dose of Toripalimab. Toripalimab (240mg dose every 3 weeks for 7 cycles, one cycle is three weeks ) will be administered as an intravenous infusion over 60 minutes.
  Interventions: Drug: Tolipalimab; Radiation: Reirradiation

INTERVENTIONS:
Drug: Tolipalimab — Radiation begun the day after the first dose of Toripalimab. Toripalimab (240mg dose every 3 weeks for 7 cycles, one cycle is three weeks) will be administered as an intravenous infusion over 60 minutes.
  Other Names: JS001
Radiation: Reirradiation — intensity-modulated radiation therapy (IMRT), 60 Gy 2.2Gy per fraction ,5 fractions per week, for 6 weeks

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of intensity-modulated radiation therapy combined with toripalimab in patients with the unresectable locally recurrent nasopharyngeal carcinoma.

DETAILED DESCRIPTION:
This is an open-label ,single center ,non-randomized, single arm exploratory study. All eligible patients presented with non-keratinizing NPC and stage rT0-4N1-3M0 /rT2-4N0M0 are assigned to receive IMRT combined with toripalimab.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed Recurrent Nasopharyngeal Carcinoma ( the recurrence time was more than 12 months from the end of the first course of radiotherapy)
2. Patients with histologically confirmed nasopharyngeal carcinoma(WHO type II-III)
3. Subjects must have measurable disease by CT or MRI per RECIST 1.1 criteria;
4. Can provide either a newly obtained or archival tumor tissue sample.
5. Tumor staged as rT0-4N1-3M0 or T2-4N0M0，II-IVa (according to the 8th AJCC edition).
6. 18 Years to 65 Years
7. Eastern Cooperative Oncology Group performance status ≤1
8. Adequate marrow function: neutrocyte count≥1.5×10e9/L, hemoglobin ≥90g/L and platelet count ≥100×10e9/L.Alanine Aminotransferase (ALT)/Aspartate Aminotransferase (AST) ≤2.5×upper limit of normal (ULN), and bilirubin ≤ 1.5×ULN. Adequate renal function: creatinine clearance rate ≥ 60 ml/min (Cockcroft-Gault formula).
9. Life expectancy ≥ 3months
10. Subjects must be willing to participate in the research and sign an informed consent form (ICF)
11. Female of child bearing potential, a negative urine or serum pregnancy test result within 72 h before study treatment. Participants of reproductive potential must be willing to use adequate contraception for the course of the study through 60 days after the last dose of Toripalimab.
12. Male subjects with WOCBP partner must be willing to use adequate contraception for the course of the study through 120 days after the last dose of Toripalimab.

Exclusion Criteria:

1. operable recurrence of nasopharyngeal cancer: rT1N0M0 rT2N0M0 (the tumour was confined in the superficial parapharyngeal spacer) rT3N0M0 (the tumour was confined in the base wall of the sphenoid sinus) rT0N1-3M0 (the tumour was not invasion into the cervical vertebrae, brachial plexus, deep muscles of the neck, or carotid artery)
2. Has known allergy to large molecule protein products or any compound of study therapy
3. Has known Subjects with other malignant tumors
4. Has any active autoimmune disease or history of autoimmune disease
5. Has a history of psychiatric substance abuse, alcoholism, or drug addiction;
6. the laboratory examination value does not meet the relevant standards within 7 days before enrollment
7. Received a systematic Glucocorticoid therapy within 4 weeks of the first dose of study medication.
8. Has a known history of active TB (bacillus tuberculosis) within 1 year; patients with adequately treated active TB with 1 year.
9. Prior therapy with a PD-1, anti-PD-Ligand 1 (PD-L1) or CTLA-4 agent;
10. Has active autoimmune disease (e.g., uveitis, enteritis, hepatitis, hypophysitis, nephritis, vasculitis, hyperthyroidism, and asthma requiring bronchodilator therapy) Patients with skin disease that doesn't require systemic treatment (e.g., vitiligo, psoriasis, or alopecia) will be allowed to enroll.
11. Has a known history of human immunodeficiency virus (HIV).
12. Has hepatitis B surface antigen (HBsAg) positive or hepatitis C virus (HCV) antibody positive
13. Has received a live vaccine within 4 weeks of planned start of study therapy
14. Pregnancy or breast feeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2023-02-01 (Estimated)

PRIMARY OUTCOMES:
ORR | Through study completion, an average of 1 year
  Objective Response Rate

SECONDARY OUTCOMES:
PFS | up to 3 years
  Progression-Free Survival is defined as time interval from recruitment to tumor progression or censoring.
OS | up to 3 years
  Overall Survival is defined as time interval from recruitment to all-caused death or censoring.
Incidence of Treatment-Emergent Adverse Events | Through study completion, an average of half a year
  Adverse events (AE), Serious Adverse Event(SAE)

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Yuan Chen, MD,PhD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Hua Y, You R, Wang Z, Huang P, Lin M, Ouyang Y, Xie Y, Zou X, Liu Y, Duan C, Liu Y, Gu C, Liu R, Yang Q, Jiang R, Zhang M, Ding X, Chen S, Lin C, Sun R, Chen M. Toripalimab plus intensity-modulated radiotherapy for recurrent nasopharyngeal carcinoma: an open-label single-arm, phase II trial. J Immunother Cancer. 2021 Nov;9(11):e003290. doi: 10.1136/jitc-2021-003290. PMID 34782428